CLINICAL TRIAL: NCT03594864
Title: Short and Long-term Outcomes After Transplantation With Hyper-reduced Liver Grafts in Low-Weight Pediatric Recipients
Brief Title: Outcomes of Liver Transplantation in Low Weight Children After Reducing the Lateral Segment of a Living Donor, Adapting the Shape and Size of the Graft to the Needs of the Recipient
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MICAELA RAICES, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 321654
Record Dates: First submitted 2018-06-16; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplantation; Low-weight Children; Hyper-reduced Liver Grafts
Keywords: Liver; Transplantation; Hyper-reduction; Graft survival; Overall survival
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hyper-reduced liver recipients.: Low-weight children who underwent live donor liver transplantation with ultrasound-guided in situ left lateral segment graft hyper-reduction.
  Interventions: Procedure: Liver transplantation with hyper-reduced grafts

INTERVENTIONS:
Procedure: Liver transplantation with hyper-reduced grafts — Live donor liver transplantation using non-anatomical in-situ ultrasound-guided reduction of left lateral segments with preparation of a graft that is larger than a monosegment, but smaller than Segments 2 and 3.

SUMMARY:
The shortage of organs has always been a problem in pediatric liver transplants due to the lack of donors with an adequate size. Different techniques of hepatic reduction have been described that allow to use larger organs in the pediatric population. However, in these techniques the maximum reduction achieved by segments 2 and 3 is excessive for low-weight children. Since 1997 the liver transplantation group at Hospital Italiano de Buenos Aires has developed and practiced a technique called hepatic hyper-reduction, which consists in reducing the lateral segment of a living donor, adapting the shape and size of the graft to the needs of the recipient. The investigators have performed approximately 50 pediatric liver transplants with live donors in low weight children in whom the hyper-reduction technique has been applied. The aim of the present study is to describe postoperative morbidity and mortality and analyze overall and graft survival.

ELIGIBILITY:
Inclusion Criteria:

* < or = 17 years old.
* Having undergone live donor liver transplantation.
* Having received hyper-reduced liver grafts
* At the Liver Transplantation Unit of the Hospital Italiano de Buenos Aires
* Between June 1997 and April 2018

Exclusion Criteria:

* > 17 years old.
* Cadaveric liver transplant
* Whole liver grafts.

Ages: 5 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients undergoing living donor liver transplantation with hyper-reduced liver grafts at the Liver Transplantation Unit of the Hospital Italiano de Buenos Aires between June 1997 and April 2018
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2018-06-03 (Actual); Study Completion 2018-06-03 (Actual)

PRIMARY OUTCOMES:
Overall survival at 1 year. | Overall survival wil be reported at 1 year after liver transplantation.
  Overall survival was defined as the time from surgery to death (all causes) or date of last follow-up, measured in months.
Overall survival at 3 years. | Overall survival wil be reported at 3 years after liver transplantation.
  Overall survival was defined as the time from surgery to death (all causes) or date of last follow-up, measured in months.
Overall survival at 10 years. | Overall survival wil be reported at 10 years after liver transplantation.
  Overall survival was defined as the time from surgery to death (all causes) or date of last follow-up, measured in months.
Graft survival at 1 year. | Graft survival wil be reported at 1 year after liver transplantation.
  Graft survival was defined as the time from surgery to the date of re-transplantation or re-entry to waiting list, measured in months.
Graft survival at 3 years. | Graft survival wil be reported at 3 years after liver transplantation.
  Graft survival was defined as the time from surgery to the date of re-transplantation or re-entry to waiting list, measured in months.
Graft survival at 10 years. | Graft survival wil be reported at 10 years after liver transplantation.
  Graft survival was defined as the time from surgery to the date of re-transplantation or re-entry to waiting list, measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Micaela Raices, Physician, Principal Investigator — Department of General Surgery, Division of HPB Surgery and Liver Transplant Unit, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Matias E Czerwonko, Physician, Study Chair — Department of General Surgery, Division of HPB Surgery and Liver Transplant Unit, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Victoria Ardiles, Physician, Study Chair — Department of General Surgery, Division of HPB Surgery and Liver Transplant Unit, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Gustavo Boldrini, Physician, Study Chair — Department of Pediatrics, Division of Pediatric Gastroenterology, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Daniel D'Agostino, Physician, Study Chair — Department of Pediatrics, Division of Pediatric Gastroenterology, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; José Marcó del Pont, Physician, Study Chair — Department of Pediatrics, Division of Pediatric Infectious Diseases, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Juan Pekolj, Doctor, Study Chair — Department of General Surgery, Division of HPB Surgery and Liver Transplant Unit, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Eduardo de Santibañes, Doctor, Study Chair — Department of General Surgery, Division of HPB Surgery and Liver Transplant Unit, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.; Martin de Santibañes, Physician, Study Director — Department of General Surgery, Division of HPB Surgery and Liver Transplant Unit, Hospital Italiano de Buenos Aires, Buenos Aires, Argentina.
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Argentina